CLINICAL TRIAL: NCT06118229
Title: A Prospective Observational Study to the Role and Impact of Wearable Smart Devices in Perioperative NSCLC Patients
Brief Title: A Study to Explore the Role and Impact of Wearable Smart Devices in Perioperative NSCLC Patients
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Professor, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: WISP-NSCLC
Record Dates: First submitted 2023-10-27; First posted 2023-11-07 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; Wearable Devices
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NSCLC patients wearing wearable smart devices: NSCLC patients wearing wearable smart devices while utilizing PROs for regular follow-up
  Interventions: Device: Wearable smart devices and PROs

INTERVENTIONS:
Device: Wearable smart devices and PROs — Patients wearing wearable smart devices to monitor physiological data while regularly utilizing PROs to report subjective assessments of their own health status.

SUMMARY:
The trial was designed as a single-center non-interventional prospective observational study to explore the role and impact of wearable smart devices in perioperative NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must provide voluntary consent to participate in this research and possess the capacity to sign an informed consent form.
2. Participants must be aged over 18 years.
3. Participants must have undergone pulmonary resection surgery with a postoperative pathological confirmation of primary lung cancer.

Exclusion Criteria:

1. Patient refusal to participate in this research.
2. Inability to wear wearable smart monitoring devices due to various reasons.
3. The pathological report suggests a non-small cell lung cancer (NSCLC) exclusion.
4. History of secondary lung cancer surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Continuously enroll all patients with non-small cell lung cancer, histopathologically confirmed
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative length of hospital stay | From time of surgery to time of discharge from the hospital (assessed up to 30 days)
  Postoperative Length of Stay (LOS) refers to the duration of a patient's hospitalization following surgery, typically measured from the completion of the surgical procedure to the time of patient discharge.

SECONDARY OUTCOMES:
Operative time | From time of the start of surgery to the end of surgery
  Operative time is defined as the time from the start of the surgical procedure to its completion, including anesthesia induction, surgical incision, manipulation of tissues, closure, and completion of all surgical tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxing He, M.D, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Department of Thoracic Surgery and Oncology, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China